CLINICAL TRIAL: NCT01128855
Title: A Double-blind, Escalating Dose, Randomized, Placebo-controlled Study to Assess the Pharmacokinetics, Safety and Tolerability of Single Subcutaneous Injections of GSK2402968 in Non-ambulant Subjects With Duchenne Muscular Dystrophy
Brief Title: A Double-blind, Escalating Dose, Randomized, Placebo-controlled Study Assessing PK, Safety, Tolerability in Non-ambulant DMD Subjects
Acronym: DEMAND I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114118
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Muscular Dystrophies
Keywords: Duchenne; Duchenne Muscular Dystrophy; DMD; 968
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): 3 mg/kg GSK2402968 / placebo
  Interventions: Drug: 3 mg/kg GSK2402968; Other: Placebo
- Cohort 2 (Experimental): 6 mg/kg GSK2402968 / placebo
  Interventions: Drug: 6 mg/kg GSK2402968; Other: Placebo
- Cohort 3 (Experimental): 9 mg/kg GSK2402968 / placebo
  Interventions: Drug: 9 mg/kg GSK2402968; Other: Placebo
- Cohort 4 (Experimental): 12 mg/kg GSK2402968 / placebo
  Interventions: Drug: 12 mg/kg GSK2402968; Other: Placebo

INTERVENTIONS:
Drug: 3 mg/kg GSK2402968 — Weekly subcutaneous injection
  Arms: Cohort 1
Drug: 6 mg/kg GSK2402968 — Weekly subcutaneous injection
  Arms: Cohort 2
Drug: 9 mg/kg GSK2402968 — Weekly subcutaneous injection
  Arms: Cohort 3
Drug: 12 mg/kg GSK2402968 — Weekly subcutaneous injection
  Arms: Cohort 4
Other: Placebo — Weekly Placebo

SUMMARY:
The purpose of this study is investigate the pharmacokinetics, safety and tolerability of single subcutaneous administration of GSK2402968 in non-ambulant boys with Duchenne muscular dystrophy

ELIGIBILITY:
Inclusion Criteria:

* Duchenne muscular dystrophy resulting from a mutation in the DMD gene, confirmed by a sponsor approved DNA diagnostic technique covering all DMD gene exons, including but not limited to MLPA (Multiplex Ligation-dependent Probe Amplification), CGH (Comparative Genomic Hybridisation), SCAIP (Single Condition Amplification/Internal Primer) or H-RMCA (High-Resolution Melting Curve Analysis), and correctable by treatment with GSK2402968.
* Age 9 years old or greater at Screening;
* Male;
* Non-ambulant (at least 1 year in a wheelchair) within the last 4 years;
* Life expectancy at least three years;
* Willingness and ability to comply with all protocol requirements and procedures;
* QTc <450msec (based on single or average QTc value of triplicate ECGs obtained over a brief recording period). Note: QTc may be either QTcB or QTcF, machine read or manual overread;
* Subjects must be willing to use adequate contraception (condoms or abstinence), from Screening until at least 5 months after the last dose of study drug;
* Informed assent and/or consent in writing signed by the subject and/or parent(s)/legal guardian (according to local regulations).

Exclusion Criteria:

* Any additional mutation (such as an additional missing exon for DMD) that cannot be treated with GSK2402968;
* Current or history of liver or renal disease;
* Acute illness within 4 weeks of anticipated administration of study medication, which may interfere with study assessments;
* Use of anticoagulants, antithrombotics or antiplatelet agents, previous treatment with investigational drugs, idebenone or other forms of Coenzyme Q10, within 6 months of the first administration of study medication;
* Start of glucocorticosteroids within 6 months or non-stable use of glucocorticosteroids within 3 months of the anticipated first administration of study medication;
* Positive hepatitis B surface antigen (HbsAg), hepatitis C antibody test (HCV), or human immunodeficiency virus (HIV) test at Screening;
* Symptomatic cardiomyopathy;
* Use of alcohol from Screening through to the 1 month Follow-up visit ;
* Any Child in Care.

Min Age: 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07-12 (Actual); Primary Completion 2011-10-25 (Actual); Study Completion 2011-10-25 (Actual)

PRIMARY OUTCOMES:
Primary Pharmacokinetic Variables:AUC, Cmax,t-max, CL/F | 35 days
Incidence of Adverse Events | 35 days
Incidence of Injection Site Reactions | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Columbus, Ohio, United States
- GSK Investigational Site, Paris, France

REFERENCES:
- See also: Results for study 114118 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114118?search=study&study_ids=114118#rs